CLINICAL TRIAL: NCT04993651
Title: Effect of Continuous Positive Airway Pressure on Fetal pH at Time of Scheduled Cesarean Delivery in Morbidly Obese Women
Brief Title: Effect of CPAP on Fetal pH at Scheduled C-section in Morbidly Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Virginia Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CPAP on Fetal pH
Record Dates: First submitted 2021-06-21; First posted 2021-08-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Morbid Obesity; Cesarean Delivery Affecting Fetus
Keywords: Fetal pH; CPAP; Continuous Positive Airway Pressure
MeSH Terms: conditions — Obesity, Morbid | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Continuous Positive Airway Pressure (Experimental): Those randomized to CPAP will be fitted with CPAP face mask or nasal device by the respiratory therapist and permitted to trial the machine to ensure proper use and fit. CPAP settings: CPAP AUTO 5-20 cm H20 will be utilized. The CPAP device will then be removed. The subject will then be placed in the supine position with a standard roll placed under the right maternal hip. Those randomized to CPAP will have the device applied and machine turned on. For those randomized to routine airway management, nasal cannula with oxygen 2L/min will be applied and this will be titrated to achieve a maternal SpO2 > 95%. End tidal CO2 monitors will be applied to both patient groups.
  Interventions: Device: CPAP
- Nasal Cannula (No Intervention): For those randomized to routine airway management, nasal cannula with oxygen 2L/min will be applied and this will be titrated to achieve a maternal SpO2 > 95%. End tidal CO2 monitors will be applied to both patient groups.

INTERVENTIONS:
Device: CPAP — CPAP is a form of noninvasive positive pressure ventilation (NPPV). CPAP works to maintain adequate levels of PO2 and PCO2 through improved alveolar ventilation and maintenance of upper-airway patency.
  Other Names: Continuous Positive Airway Pressure
  Arms: Continuous Positive Airway Pressure

SUMMARY:
The objective of our study is to evaluate the effect of CPAP on umbilical cord acid base status in morbidly obese women at the time of scheduled cesarean delivery. We hypothesize that neonates born to mothers wearing CPAP during the cesarean section will have a higher umbilical artery pH.

DETAILED DESCRIPTION:
This is a randomized control trial comparing CPAP to routine airway management in morbidly obese patients undergoing scheduled cesarean delivery. Morbidly obese women meeting criteria for inclusion will be approached for participation. Women who are scheduled for cesarean delivery at Sentara Norfolk General Hospital will be approached at a prenatal appointment prior to scheduled date of delivery. If a woman agrees to participate in the study, she will be counseled and consented at that time.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between the ages of 18-45
* Body mass index of 40 kg/m2 or greater at the time patient is scheduled for cesarean delivery
* Singleton gestation
* Scheduled for primary or repeat cesarean delivery at Sentara Norfolk General Hospital
* Gestational age between 37+0 and 41+0 weeks at the time of delivery
* Non-stress test on admission with moderate variability, without repetitive late or variable decelerations
* Negative SARS-CoV-2 PCR test within 72 hours of procedure

Exclusion Criteria:

* Fetal growth restriction
* Active pulmonary diseases to include pneumonia, sarcoidosis, pulmonary hypertension, moderate or severe persistent asthma
* Suspected placenta accreta based on prenatal sonographic evaluation
* Active maternal infection to include pyelonephritis, appendicitis, upper respiratory tract infection, urinary tract infection or suspected intra-amniotic infection
* SARS-CoV-2 positive test within past 10 days or ongoing symptoms of SARS-CoV-2 to include cough, fever or shortness of breath with positive test greater than 10 days prior, or history of hospitalization for SARS-CoV-2 infection
* Fetus with aneuploidy or major anomaly
* Enrolled in another trial that may affect outcome

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Umbilical Cord Arterial pH | At delivery
  We hypothesize that neonates born to mothers wearing CPAP during the cesarean section will have a higher umbilical artery pH.

SECONDARY OUTCOMES:
Patient satisfaction with use of CPAP | Within 4 days following delivery (prior to discharge from hospital)
  Survey will be used to determine patient experience and satisfaction
Effect of CPAP on maternal acid base status with analysis of venous blood gas | At time of uterine incision
  Maternal venous blood gas will be analyzed at the time of uterine incision to measure the acid base status
Effect of maternal CPAP use on neonatal Apgar scores | At delivery
  Apgar scores will be compared between 2 groups
Effect of maternal CPAP use on composite neonatal outcome | At delivery
  Perinatal death, respiratory support, Apgar score <=3 at 5 min, hypoxic ischemic encephalopathy, hypotension requiring vasopressor support
Effect of duration in supine position prior to delivery on neonatal acid base status | At delivery
  Neonatal venous blood gas will be analyzed to determine the acid base status as it correlates to length of time in maternal supine position
Effect of duration in supine position prior to delivery on maternal acid base status | At delivery
  Maternal venous blood gas will be analyzed to determine the acid base status as it correlates to length of time in supine position

CONTACTS AND LOCATIONS:
Overall Officials: Tracey DeYoung, MD, Principal Investigator — Eastern Virginia Medical School
Locations (1):
- Department of Obstetrics and Gynecology, Division of Maternal-Fetal Medicine, Eastern Virginia Medical School, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Flegal KM, Kruszon-Moran D, Carroll MD, Fryar CD, Ogden CL. Trends in Obesity Among Adults in the United States, 2005 to 2014. JAMA. 2016 Jun 7;315(21):2284-91. doi: 10.1001/jama.2016.6458. PMID 27272580
- [Background] Chu SY, Kim SY, Schmid CH, Dietz PM, Callaghan WM, Lau J, Curtis KM. Maternal obesity and risk of cesarean delivery: a meta-analysis. Obes Rev. 2007 Sep;8(5):385-94. doi: 10.1111/j.1467-789X.2007.00397.x. PMID 17716296
- [Background] Weiss JL, Malone FD, Emig D, Ball RH, Nyberg DA, Comstock CH, Saade G, Eddleman K, Carter SM, Craigo SD, Carr SR, D'Alton ME; FASTER Research Consortium. Obesity, obstetric complications and cesarean delivery rate--a population-based screening study. Am J Obstet Gynecol. 2004 Apr;190(4):1091-7. doi: 10.1016/j.ajog.2003.09.058. PMID 15118648
- [Background] Hibbard JU, Gilbert S, Landon MB, Hauth JC, Leveno KJ, Spong CY, Varner MW, Caritis SN, Harper M, Wapner RJ, Sorokin Y, Miodovnik M, Carpenter M, Peaceman AM, O'Sullivan MJ, Sibai BM, Langer O, Thorp JM, Ramin SM, Mercer BM, Gabbe SG; National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Trial of labor or repeat cesarean delivery in women with morbid obesity and previous cesarean delivery. Obstet Gynecol. 2006 Jul;108(1):125-33. doi: 10.1097/01.AOG.0000223871.69852.31. PMID 16816066
- [Background] Edwards RK, Cantu J, Cliver S, Biggio JR Jr, Owen J, Tita ATN. The association of maternal obesity with fetal pH and base deficit at cesarean delivery. Obstet Gynecol. 2013 Aug;122(2 Pt 1):262-267. doi: 10.1097/AOG.0b013e31829b1e62. PMID 23969793
- [Background] Vricella LK, Louis JM, Mercer BM, Bolden N. Impact of morbid obesity on epidural anesthesia complications in labor. Am J Obstet Gynecol. 2011 Oct;205(4):370.e1-6. doi: 10.1016/j.ajog.2011.06.085. Epub 2011 Jun 29. PMID 21864821
- [Background] von Ungern-Sternberg BS, Regli A, Bucher E, Reber A, Schneider MC. Impact of spinal anaesthesia and obesity on maternal respiratory function during elective Caesarean section. Anaesthesia. 2004 Aug;59(8):743-9. doi: 10.1111/j.1365-2044.2004.03832.x. PMID 15270963
- [Background] Kelly MC, Fitzpatrick KT, Hill DA. Respiratory effects of spinal anaesthesia for caesarean section. Anaesthesia. 1996 Dec;51(12):1120-2. doi: 10.1111/j.1365-2044.1996.tb15046.x. PMID 9038445
- [Background] Turan OM, Rosenbloom J, Galey JL, Kahntroff SL, Bharadwaj S, Turner SM, Malinow AM. The Relationship between Rostral Retraction of the Pannus and Outcomes at Cesarean Section. Am J Perinatol. 2016 Aug;33(10):951-6. doi: 10.1055/s-0036-1581054. Epub 2016 Apr 21. PMID 27100522
- [Background] Dominguez JE, Krystal AD, Habib AS. Obstructive Sleep Apnea in Pregnant Women: A Review of Pregnancy Outcomes and an Approach to Management. Anesth Analg. 2018 Nov;127(5):1167-1177. doi: 10.1213/ANE.0000000000003335. PMID 29649034
- [Background] Dominguez JE, Street L, Louis J. Management of Obstructive Sleep Apnea in Pregnancy. Obstet Gynecol Clin North Am. 2018 Jun;45(2):233-247. doi: 10.1016/j.ogc.2018.01.001. PMID 29747728
- [Background] MacIntyre NR. Physiologic Effects of Noninvasive Ventilation. Respir Care. 2019 Jun;64(6):617-628. doi: 10.4187/respcare.06635. PMID 31110031
- [Background] Corcione N, Karim H, Mina B, Pisano A, Dikmen Y, Kondili E, Nicolini A, Fiorentino G, Caldeira V, Ubeda A, Papadakos P, Wittenstein J, Singha S, Sovani M, Panda C, Tani C, Khatib M, Perren A, Ho K, Esquinas A. Non-invasive ventilation during surgery under neuraxial anaesthesia: a pathophysiological perspective on application and benefits and a systematic literature review. Anaesthesiol Intensive Ther. 2019;51(4):289-298. doi: 10.5114/ait.2019.88572. PMID 31617693
- [Background] Erdogan G, Okyay DZ, Yurtlu S, Hanci V, Ayoglu H, Koksal B, Turan IO. Non-invasive mechanical ventilation with spinal anesthesia for cesarean delivery. Int J Obstet Anesth. 2010 Oct;19(4):438-40. doi: 10.1016/j.ijoa.2010.04.005. Epub 2010 Aug 10. PMID 20702082
- [Background] Polin CM, Hale B, Mauritz AA, Habib AS, Jones CA, Strouch ZY, Dominguez JE. Anesthetic management of super-morbidly obese parturients for cesarean delivery with a double neuraxial catheter technique: a case series. Int J Obstet Anesth. 2015 Aug;24(3):276-80. doi: 10.1016/j.ijoa.2015.04.001. Epub 2015 Apr 8. PMID 25936783
- [Background] Chung F, Yang Y, Liao P. Predictive performance of the STOP-Bang score for identifying obstructive sleep apnea in obese patients. Obes Surg. 2013 Dec;23(12):2050-7. doi: 10.1007/s11695-013-1006-z. PMID 23771818
- [Background] Pearson F, Batterham AM, Cope S. The STOP-Bang Questionnaire as a Screening Tool for Obstructive Sleep Apnea in Pregnancy. J Clin Sleep Med. 2019 May 15;15(5):705-710. doi: 10.5664/jcsm.7754. PMID 31053210
- [Background] Simon VB, Fong A, Nageotte MP. Supplemental Oxygen Study: A Randomized Controlled Study on the Effect of Maternal Oxygen Supplementation during Planned Cesarean Delivery on Umbilical Cord Gases. Am J Perinatol. 2018 Jan;35(1):84-89. doi: 10.1055/s-0037-1606184. Epub 2017 Aug 24. PMID 28838010
- [Background] Skiold B, Petersson G, Ahlberg M, Stephansson O, Johansson S. Population-based reference curve for umbilical cord arterial pH in infants born at 28 to 42 weeks. J Perinatol. 2017 Mar;37(3):254-259. doi: 10.1038/jp.2016.207. Epub 2016 Dec 1. PMID 27906196
- [Background] Johansson S, Sandstrom A, Cnattingius S. Maternal overweight and obesity increase the risk of fetal acidosis during labor. J Perinatol. 2018 Sep;38(9):1144-1150. doi: 10.1038/s41372-018-0144-5. Epub 2018 Jun 19. PMID 29915374